CLINICAL TRIAL: NCT01580553
Title: The Clinical Study of the Efficacy and Safety of L-Carnitine Injection in Treatment of Heart Failure -A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: The Clinical Study of the Efficacy and Safety of L-Carnitine Injection in Treatment of Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LeesPharm_LC-HF
Record Dates: First submitted 2012-03-28; First posted 2012-04-19 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Heart Failure,
Keywords: Heart failure; L-carnitine; injection; safety; efficacy
MeSH Terms: conditions — Heart Failure | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levocarnitine (Placebo Comparator)
  Interventions: Drug: Levocarnitine placebo
- L-carnitine (Active Comparator)
  Interventions: Drug: Levocarnitine Injection

INTERVENTIONS:
Drug: Levocarnitine Injection — Levocarnitine Injection:5ml:1g
  Arms: L-carnitine
Drug: Levocarnitine placebo — L-Carnitine injection placebo (5ml:1g)
  Arms: Levocarnitine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of L-carnitine injection in treatment of Chinese patients with heart failure.

A prospective, multicenter, randomized, double-blind, parallel, placebo-controlled clinical study was performed.

Treatment period: 7 days, follow-up: 1 month

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy and safety of L-carnitine injection in treatment of Chinese patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. The subject aged ≥ 18 years, men or women.
2. The subject has a diagnosis of chronic left heart or right heart failure (a past medical history of left heart failure caused by coronary heart disease, hypertension and dilated cardiomyopathy, or a medical history of right heart failure caused by pulmonary artery hypertension (the 1st type of diagnostic classification, WHO conference, Venice, 2003) and left heart disease (the 2nd type) ;the case number of right heart failure is about 30% of the total case number).
3. The subject needs hospitalization because of heart failure and will stay in hospital for more than 7 days.
4. NYHA-FC is Class II- IV (Class II cases < 20%, except the refractory terminal heart failure patients).
5. The subject's UCG shows that LVEF ≤ 45％ (left heart failure).
6. CI < 2.5 L/min/m2 or CO < 4L/min (right heart failure)
7. The subject has signed the ICF.

Exclusion Criteria:

1. Subjects with medical history of heart failure caused by valvular heart disease, mechanical obstruction, pericardial disease and myocardial amyloidosis.
2. Subjects with heart function Class IV that have unstable hemodynamics and need final stage cardiac transplantation and intravenous vasoactive drugs.
3. Subjects will leave the hospital in 7 days.
4. Subjects with severe cerebral apoplexy (life threatening).
5. Subjects with AMI or acute pulmonary embolism.
6. Subjects with uremia and did not undergo dialysis.
7. Subjects with COPD.
8. Subjects with severe anemia (Hb≤60g/l).
9. Subject who is receiving other metabolism improving drugs within one month (such as trimetazidine dihydrochloride tablets and 1, 6- fructose diphosphate.
10. Subject with other severe disease and his/her life expectancy <12 months.
11. Subject who has participated in other clinical trial within 3 months or is participating in other study.
12. Subject who has received L-carnitine treatment within 1 month.
13. Subject who is allergic to L-carnitine and its derivatives.
14. Subject is receiving other cardiotoxic drugs.
15. Subjects with medical history of epilepsy.
16. Subject who is a drug or alcohol abuser.
17. Subject who has received PCI, CABG or vascular remodeling.
18. Subject with arrhythmia that the investigator thinks unsuitable to include.
19. The subject who is pregnant or lactating, and the woman of childbearing age has not taken contraception measures.
20. The subject has not signed the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
NYHA cardiac functional grading | 7 days treatment
  The cardiac functional changes between the end of medication (within 24 hrs) and baseline (prior to medication) are evaluated by the three-grade criteria (excellent, effective and no response). And calculate the effective rate.
  Excellent: cardiac function improved for 2 grades and above Effective: cardiac function improved for one grade No response: failed to achieve the effective criteria.

SECONDARY OUTCOMES:
Other efficacy evaluations | 7 days treatment
  6-Minute Walk Test (6MWT)
Other efficacy evaluations | 7 days treatment
  2.Incidence of major cardiovascular events when follow-up (within 1 month)
  * symptoms get worse (NYHA cardiac functional grading aggravates)
  * increase dosage or other treatment for aggravating heart failure
  * need hospitalization again for heart failure or other reasons
  * death
Other efficacy evaluations | 7 days treatment
  Plasma L-carnitine level (acyl-carnitine/free carnitine)
Other efficacy evaluations | 7 days treatment
  ultrasound echocardiography to measure left ventricular ejection fraction (LVEF)
Other efficacy evaluations | 7 days treatment
  measure the N-Terminal-pro brain natriuretic peptide level in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital affiliated to Tongji University, Shanghai, China